CLINICAL TRIAL: NCT00328471
Title: A Post Discharge Intervention to Improve Stroke Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Dr. Kyle Allen, Summa Health system
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R01NS041333-01A1 (NIH); 1R01NS041333-01A1 (NIH)
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Cerebrovascular Accident
Keywords: patient care management; cerebrovascular accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: care management

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to test the effectiveness of a comprehensive interdisciplinary post-discharge stroke care management intervention in improving the overall well-being of 190 stroke survivors as compared to 190 patients who receive usual post-discharge stroke care.

DETAILED DESCRIPTION:
The major components of the model of post-stroke care being tested include equal emphasis on physical and psychosocial issues known to impact stroke outcomes, an Advanced Practice Nurse care manager (APN-CM), an interdisciplinary healthcare team, evidenced-based care plans, collaboration with the patient's primary care physician (PCP), and ongoing patient monitoring. The APN-CM will work as part of an interdisciplinary post-stroke consultation team (PSC-Team) that will review problems identified at an in-home patient assessment. The core PSC-Team will include a geriatrician, a community-based general internist, a Clinical Nurse Specialist from the acute stroke unit, the APN-CM, and a physical therapist. Extended team members will be available as-needed and will include a neurologist, pharmacist, physiatrist, social worker, speech therapist, occupational therapist, and dietitian. The PSC-Team will develop patient care plans specific to each problem identified by the APN-CM. A copy of the care plans, evidence-based guidelines, pertinent references, and a short paragraph providing "academic detailing" specific to the patient's problems will be given to the patient's PCP by phone and in writing. The APN-CM will work collaboratively with the PCP to implement the recommendations and provide ongoing monitoring.The primary outcome of overall well-being of stroke survivors will be obtained at 6 months.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of ischemic stroke. NIH Stroke Scale score >1. Discharged to home from the acute care hospital, or discharged to home within 4 weeks from a short term skilled nursing facility (SNF) or acute rehabilitation facility.

Live within 25 miles of the study site. English speaking. Do not have an endarterectomy planned at the time of discharge to home.

Exclusion Criteria:

Has other illness that would dominate post-stroke care (e.g., terminal diagnosis, dialysis patient, severe dementia/Alzheimer's disease).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2002-06; Primary Completion 2008-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle R Allen, DO, Principal Investigator — Summa Health System

REFERENCES:
- [Result] Allen KR, Hazelett SE, Palmer RR, Jarjoura DG, Wickstrom GC, Weinhardt JA, Lada R, Holder CM, Counsell SR. Developing a stroke unit using the acute care for elders intervention and model of care. J Am Geriatr Soc. 2003 Nov;51(11):1660-7. doi: 10.1046/j.1532-5415.2003.51521.x. PMID 14687400
- [Result] Allen KR, Hazelett S, Jarjoura D, Wickstrom GC, Hua K, Weinhardt J, Wright K. Effectiveness of a postdischarge care management model for stroke and transient ischemic attack: a randomized trial. J Stroke Cerebrovasc Dis. 2002 Mar-Apr;11(2):88-98. doi: 10.1053/jscd.2002.127106. PMID 17903862
- [Result] Allen KR, Hazelett SE, Jarjoura DG, Wright K, Clough L, Weinhardt J. Improving stroke outcomes: implementation of a postdischarge care management model. Journal of clinical outocmes management 11(11):707-714,2004.